CLINICAL TRIAL: NCT00881829
Title: Accuracy Validation in Multiple SpO2 Systems
Brief Title: Hypoxia Blood Validation in Multiple Pulse Oximeters
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clinimark, LLC (Other)
Responsible Party: Principal Investigator, David Ransom, MD, Primary Investigator, Clinimark, Clinimark, LLC
Other Study IDs: PR 2016-192 Rev 1
Record Dates: First submitted 2009-04-13; First posted 2009-04-15 (Estimated); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Hypoxia
Keywords: Pulse Oximetry; Temperature; Respiratory Rate; Respiratory Gases; This study determine the measurement accuracy of the physiological parameters
MeSH Terms: conditions — Hypoxia | interventions — Blood Pressure; Respiratory Rate; Body Temperature

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Healthy volunteer: Smoker or non-smoker
  Interventions: Device: Pulse Oximeter, Blood Pressure, Respiratory Rate, Respiratory Gasses, Temperature

INTERVENTIONS:
Device: Pulse Oximeter, Blood Pressure, Respiratory Rate, Respiratory Gasses, Temperature — Measurement of physiological parameters.

SUMMARY:
The purpose of this study is to evaluate the SpO2 accuracy and performance of multiple pulse oximeters during non-motion conditions over the range of 70-100% SaO2 as compared to arterial blood samples assessed by CO-Oximetry for SpO2 validation.

This study is observational in nature which quantifies device performance and accuracy in comparison to a Reference Standard.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the SpO2 accuracy and performance of pulse oximeters during non-motion conditions over the range of 70-100% SaO2 as compared to arterial blood samples assessed by CO-Oximetry for SpO2 validation. The end goal is to show the SpO2 accuracy performance of the pulse oximeters. It is expected that the Accuracy Root Mean Square (Arms) performance of pulse oximeters will meet a specification of 3 or better in non-motion conditions for the range of 70-100% SaO2 thereby demonstrating an acceptable SpO2 accuracy performance specification

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals between the age of 18-50 years.

Exclusion Criteria:

* Clotting disorders, diabetes, currently taking psychotropic medications.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Residents of the Denver metropolitan area.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-08-09 (Actual); Primary Completion 2021-12-21 (Estimated); Study Completion 2021-12-21 (Estimated)

PRIMARY OUTCOMES:
Completion of study by all subjects | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: David Ransom, MD, Principal Investigator — Avista Adventist Hospital
Locations (1):
- Clinimark Laboratories, Louisville, Colorado, United States